CLINICAL TRIAL: NCT01357824
Title: View af Larynx and Intubation With a Flexible Fibreoptic Scope With and Without Sellick´s Maneuver.
Brief Title: Fibreoptic Intubation With and Without Sellick´s Maneuver
Status: Completed | Type: Observational
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Bjorn Arenkiel, Reservelæge, Glostrup University Hospital, Copenhagen
Other Study IDs: Glostrup Crich Study
Record Dates: First submitted 2011-05-19; First posted 2011-05-23 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Intubation Intraesophageal; Respiratory Aspiration of Gastric Contents
Keywords: Intubation; Sellick´s maneuver; aspiration; [E05.497.578]
MeSH Terms: conditions — Respiratory Aspiration of Gastric Contents

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients admitted for elective surgery: The patient admitted for elective surgery can be included, and will both the case and control, as we intubate the same patient twice, with and without Sellick´s maneuver.
  Interventions: Procedure: Application of Sellick´s maneuver.

INTERVENTIONS:
Procedure: Application of Sellick´s maneuver. — The patient will be intubated with a flexible fiberscope, Olympus model, under the application of Sellick´s maneuver, with the recommended 30 Newtons pressure, and also, as control, be intubated with a sham Sellick´s maneuver, with 0 Newton. The order of the pressures is randomized, and it is blinded to the intubating physician by a cloth which of the maneuvers that is used. The pressure is measured be a pediatric cuff, which is pressed against the throat.

SUMMARY:
The goal of this study is to evaluate the effect of Sellick´s Maneuver, a firm pressure on the throat, just below the Adams apple, to occlude the esophagus, in order to prevent aspiration of gastric contents, on intubation with a flexible fiberscope. The result of this study will be participate in the discussion of the importance of Sellick´s Maneuver.

DETAILED DESCRIPTION:
The patients included in this study has volunteered after sufficient information, and must be ASA-class I-II, 18 years or more, and must not have indications for a rapid sequence induction.

The patient will be intubated twice, with and without Sellick´s maneuver. It is blinded to the intubating physician, in which order this pressure is applied.

The outcomes measures will be time of intubation, oxygen saturation before and after intubation and a Cormack Scale graduation of the visibility of the vocal cords. The intubation will be failed, if it cannot be performed under 120 seconds, or if the patients desaturate to 95% or less.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Informed consent to participate in the study
* Age 18 or older
* Predicted difficult airways

Exclusion Criteria:

* Body mass index more then 35
* Patients with an indication for a rapid sequence induction (reflux, Hiatus herniation, Gastric bypass)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted for elective surgery at Glostrup University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Time of intubation | 180 seconds
  The investigators will find an eventually change in the time of intubation with and without Sellick´s Maneuver

SECONDARY OUTCOMES:
Number of patients that cannot be intubated after 120 sec. with and without Sellick´s maneuver | 180 seconds
  Patients that is not intubated after 120 seconds in each trial, will count as "not intubated after 120 seconds".
Fall of oxygen saturation after intubation with and without Sellick´s maneuver. | 180 seconds
  The investigators measure the oxygen saturation on a finger device at the beginning and the and of the intubations.
Visualization of the vocal cords | 180 seconds
  The investigators will observe the visualization of the vocal cords, and provide the result on the Cormack Score.

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn Arenkiel, MD, Principal Investigator — Glostrup University Hospital, Copenhagen
Locations (1):
- Operations- og Anæstesilogisk afd Y, Glostrup Hospital, Glostrup Municipality, Denmark

REFERENCES:
- [Background] Smith CE, Boyer D. Cricoid pressure decreases ease of tracheal intubation using fibreoptic laryngoscopy (WuScope System. Can J Anaesth. 2002 Jun-Jul;49(6):614-9. doi: 10.1007/BF03017391. PMID 12067876
- [Background] Asai T, Goy RW, Liu EH. Cricoid pressure prevents placement of the laryngeal tube and laryngeal tube-suction II. Br J Anaesth. 2007 Aug;99(2):282-5. doi: 10.1093/bja/aem159. Epub 2007 Jun 15. PMID 17573388
- [Background] Haslam N, Parker L, Duggan JE. Effect of cricoid pressure on the view at laryngoscopy. Anaesthesia. 2005 Jan;60(1):41-7. doi: 10.1111/j.1365-2044.2004.04010.x. PMID 15601271
- [Background] Brisson P, Brisson M. Variable application and misapplication of cricoid pressure. J Trauma. 2010 Nov;69(5):1182-4. doi: 10.1097/TA.0b013e3181d2793e. PMID 21068621
- [Background] Ellis DY, Harris T, Zideman D. Cricoid pressure in emergency department rapid sequence tracheal intubations: a risk-benefit analysis. Ann Emerg Med. 2007 Dec;50(6):653-65. doi: 10.1016/j.annemergmed.2007.05.006. Epub 2007 Aug 3. PMID 17681642
- [Background] Priebe HJ. Cricoid pressure: an expert's opinion. Minerva Anestesiol. 2009 Dec;75(12):710-4. PMID 19940824